CLINICAL TRIAL: NCT05492422
Title: Evaluating the Efficacy of Sequenced Central Executive and Behavioral Parent Training for Children with ADHD
Brief Title: Central Executive Training and Parent Training for ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Kofler, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01MH125893 (NIH)
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- CET-then-BPT (Experimental): Families receive CET in Phase 1 followed by BPT in Phase 2
  Interventions: Device: Central Executive Training (CET); Behavioral: Behavioral Parent Training (BPT)
- BPT-then-CET (Experimental): Families receive BPT in Phase 1 followed by CET in Phase 2
  Interventions: Device: Central Executive Training (CET); Behavioral: Behavioral Parent Training (BPT)
- Waitlist then CET+BPT (Experimental): Families do not receive either intervention in Phase 1 and then receive both CET and BPT concurrently in Phase 2
  Interventions: Device: Central Executive Training (CET); Behavioral: Behavioral Parent Training (BPT)
- CET+BPT then 'waitlist' (follow-up) (Experimental): Families receive CET and BPT concurrently in Phase 1, and then are followed in Phase 2 with not additional intervention
  Interventions: Device: Central Executive Training (CET); Behavioral: Behavioral Parent Training (BPT)

INTERVENTIONS:
Device: Central Executive Training (CET) — Central Executive Training (CET)
Behavioral: Behavioral Parent Training (BPT) — Behavioral Parent Training (BPT)

SUMMARY:
The goal of the current project is to combine two evidence- based treatments for school-aged children with ADHD: Central Executive Training (CET) and Behavioral Parent Training (BPT). CET is a computerized training intervention that improves ADHD symptoms and academic functioning by improving children's working memory abilities. BPT is a therapeutic intervention that improves family functioning and child oppositional-defiant (ODD) symptoms by changing parenting behaviors. Their combined use is expected to provide complementary and additive benefits, particularly if CET is delivered before BPT.

ELIGIBILITY:
Inclusion:

1. Children ages 8-12 with principal ADHD diagnoses (via K-SADS); and
2. parent AND teacher ratings in clinical/borderline range based on age and sex on ADHD Rating Scale (ADHD-5) or Behavior Assessment Scale for Children (BASC-3) Attention Problems/Hyperactivity subscales (i.e., 90th percentile or higher based on both informants).

All DSM-5 ADHD presentations will be eligible.

Exclusion:

1. gross neurological, sensory, or motor impairment;
2. history of seizure disorder, psychosis, bipolar, or severe dysregulation disorders that may interfere with participation (e.g., disruptive mood dysregulation, intermittent explosive, reactive attachment, substance use);
3. intellectual disability or Wechsler Intelligence Scale for Children (WISC-V) short-form standard score <70;
4. conditions requiring acute intervention, e.g., active suicidality; and
5. non-English speaking child or parent.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Rapport visuospatial/phonological working memory test | Administered during a 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
Alabama parenting scale | Parent questionnaire requiring approximately 15 minutes to complete, administered to parent while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
Parenting sense of competence scale | Parent questionnaire requiring approximately 15 minutes to complete, administered to parent while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
Parent stress index | Parent questionnaire requiring approximately 15 minutes to complete, administered to parent while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session

SECONDARY OUTCOMES:
Behavior Assessment System for Children | Parent and teacher questionnaire requiring approximately 15 minutes to complete, administered to parent and mailed to teacher while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
ADHD Rating Scale | Parent and teacher questionnaire requiring approximately 15 minutes to complete, administered to parent and mailed to teacher while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
ODD symptoms (DSM-based checklist) | Parent and teacher questionnaire requiring approximately 15 minutes to complete, administered to parent and mailed to teacher while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session

OTHER OUTCOMES:
Academic performance rating scale | Teacher questionnaire requiring approximately 15 minutes to complete, mailed to teacher within 2 weeks of last intervention session
Parent relationship questionnaire | Parent questionnaire requiring approximately 15 minutes to complete, administered to parent while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
Dyadic parent-child interaction coding system (DPICS) | Structured parent-child interaction conducted during the post-treatment testing session within 2 weeks of final intervention session

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided